CLINICAL TRIAL: NCT06445101
Title: Vital@Work: an Evidence-based Intervention Program for Prevention of Mental Health Complaints at Work, Tailored to Specific Organisational Needs and Contextual Factors
Brief Title: Vital@Work: an Intervention for Prevention of Mental Health Complaints at Work
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Health Holland (Other); Stichting Trimbos-Instituut (Other)
Responsible Party: Principal Investigator, Luuk Bouwens, PhD Candidate, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: LSHM22035-H025
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stress
Keywords: work-related emotional exhaustion

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial comparing intervention group with care as usual group.
  Randomization is carried out at the cluster (team or department) level to prevent contamination between employees assigned to the intervention group and those in the control group.
Who Masked: Participant
Masking Description: Due to the PA intervention and associated activities, it is not possible to blind the researchers and department managers to the condition they are assigned to. However, employees in the departments randomized to the intervention or control group are not aware of the research design. Only department managers are informed about the research design and the outcome of randomization, and they are asked not to communicate the research design to the employees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participatory Approach (intervention) (Experimental): Employees in departments allocated to the intervention group receive the PA strategy in addition to the existing range of preventive mental health measures within the organization.
  Interventions: Other: Participatory Approach
- Care as usual (No Intervention): Departments assigned to the control group receive usual strategies and therefore only have access to the existing range of preventive interventions within the organization (without the PA intervention).

INTERVENTIONS:
Other: Participatory Approach — The participatory approach is a stepwise, collaborative approach to the analysis and solvation of bottlenecks that cause stress in employees.
  Arms: Participatory Approach (intervention)

SUMMARY:
The objective of the current study, Vital@Work, is to keep employees in the Netherlands vital on the long term by preventing work-related mental health problems. Therefore, we test an evidence based Participatory Approach (PA) to compose a mental health program tailored to behavioral, organizational & contextual (BOC) determinants of individuals and populations at risk. The PA is investigated in four different organizations, which differ in sector, size (small and large organizations), type of organization (private or public) and type of work. The varied organizations, each characterized by unique BOC-determinants, provide an opportunity for researching tailored intervention activities that aim to effectively prevent work-related mental health problems. By identifying common factors across these diverse organizations, we aim to grasp patterns of mechanisms for interventions to mental health at work. By doing this, we come closer to opening black box of how and why interventions work and thus closer to tailoring interventions to needs of both individuals and organizations

DETAILED DESCRIPTION:
This study evaluates the PA as a strategy to implement measures to prevent or reduce work-related mental health problems by a cluster randomized controlled trial, including an intervention and control group. Employees in departments allocated to the intervention group receive the PA intervention in addition to the existing range of preventive mental health measures within the organization. Departments assigned to the control group receive standard practice and therefore only the existing range of preventive interventions will be highlighted and further drawn to the attention of employees (without the PA intervention). Due to the PA intervention and associated activities, it is not possible to blind the researchers and department managers. However, employees in the departments randomized to the intervention or control group are not aware of the research design. Only department managers are informed about the research design and the outcome of randomization, and they are asked not to communicate the research design to the employees.

The PA consists of six steps: 1) preparation: create prerequisites and initiate the PA, 2) risk assessment: analysis of bottlenecks and risks 3) solutions: Analysis of potential solutions 4) action planning: jointly formulating a plan of action to realize solutions 5) implementation: implementing measures by means of the action plan and 6) evaluation: evaluation of the approach.

For each intervention group, a participatory working group will be established, comprising 5-7 employees, a department manager/supervisor, a health and safety coordinator, an HR representative, and a communication specialist. Each intervention group is coordinated by a process facilitator who is responsible for preparing the meetings with the working group and leading the discussions during these sessions. To prepare individuals for this role, the process facilitator receives training, provided by researchers experienced in the PA.

The participative working group will go through steps 2 to 4 of the PA during a day session, resulting in an action plan for the intervention activities to be implemented. Subsequently, this action plan will be implemented throughout the entire team comprising the intervention group. This implementation process will be led by the process facilitator, supported by change agents. Ideally, (some of) the working group members will act as change agents. Change agents have the task of implementing interventions as widely as possible within the department and ensuring a smooth implementation process so that employees actually make use of the innovations. In order to act as catalysts for the implementation process within the department, the change agents and the process facilitator are trained by researchers experienced in the PA. The duration of the entire implementation period is approximately 12 months, but depends on the selected intervention activities, with short-term implementations lasting < 3 months, and long-term implementations lasting > 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion will be done on cluster level (e.g. team or department), after discussing this with participating organizations. The inclusion criteria for participation in the study comprise being at least 18 years of age, holding an employment contract with the participating organization.

Exclusion Criteria:

* The exclusion criteria include being under 18 years old, not being part of the participating teams/departments, or not having an employment contract with the participating organization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stress | Baseline - 6 months after baseline - 12 months after baseline
  Stress will be assessed using the stress subscale of the short version of the Depression Anxiety and Stress Scale (DASS-21; Lovibond & Lovibond, 1995), designed to measure the emotional states of depression, anxiety and stress. The stress subscale of DASS-21 comprises seven statements. Participants indicate the extent to which these statements applied to them during the past week, using a Likert scale ranging from 0 ('never') to 3 ('almost always').

SECONDARY OUTCOMES:
Work related psychosocial risk factors | Baseline - 6 months after baseline - 12 months after baseline
  At the individual level, we will assess work-related psychosocial risk factors, including job demands, autonomy, supervisor support and co-worker support. For measuring job demands, we will utilize four subscales from the validated Dutch version of The Copenhagen Psychosocial Questionnaire (COPSOQ-III; Burr et al., 2019; Kristensen et al., 2005) subscales quantitative demands, cognitive demands, emotional demands and work pace. The COPSOQ is a globally recognized and extensively employed tool for assessing a range of psychosocial factors in workplaces (Burr et al., 2019)
Sense of community | Baseline - 6 months after baseline - 12 months after baseline
  Sense of Community will be measured using three items form the validated Dutch version of COPSOQ-III (Burr et al., 2019; Kristensen et al., 2005)
Psychosocial safety climate | Baseline - 6 months after baseline - 12 months after baseline
  At employee level, the Psychosocial Safety Climate (PSC) is assessed using the Dutch translation of the PSC-4, a shortened version of the PSC-12 (Dollard, 2019).
Presenteeism and absenteeism | Baseline - 6 months after baseline - 12 months after baseline
  Presenteeism will be assessed by two items of the World Health Organization Health and Work Performance Questionnaire (HPQ) (Kessler et al., 2003) and an item obtained from Vänni et al. (2018). The absenteeism history of the employee in the twelve months prior to the survey will be assessed using a set of three questions. Additionally, two questions will be included regarding the most recent absenteeism incident experienced by employees. This most recent incident may potentially have occurred more than twelve months ago, allowing for responses from employees who have not been absent in the past twelve months but were absent before that period. They are asked about the type of complaints that led to their most recent absence and whether these complaints were work-related.
Implementation outcomes | Baseline - 6 months after baseline - 12 months after baseline
  To assess implementation outcomes, a series of questions (12 items) will be used concerning existing and recently introduced resources (interventions, measures, policies, and additional support) designed to foster mental health and prevent related issues. These items focus on the availability and utilization of existing and newly provided resources.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - GGZ Ingeest, Amsterdam
  - Transavia, Amsterdam
  - RSO, The Hague

REFERENCES:
- [Derived] Bouwens L, Anema JR, Juurlink TT, Beekman ATF, Schelvis RMC. Protocol of a randomized controlled multicenter trial investigating process and effectiveness of a participatory organizational approach for preventing work-related mental health problems among employees: vital@work. BMC Public Health. 2025 Aug 30;25(1):2970. doi: 10.1186/s12889-025-24367-8. PMID 40885945